CLINICAL TRIAL: NCT02058628
Title: A Multi-centre, Single-blind, Parallel Group, Clinical Evaluation of the Efficacy and Safety of Clindamycin 1% / Benzoyl Peroxide 3% and Azelaic Acid 20% in the Topical Treatment of Mild to Moderate Acne Vulgaris
Brief Title: Comparison of the Efficacy and Safety of Clindamycin + Benzoyl Peroxide Formulation With Azelaic Acid Formulation in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200398
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Results first posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Acne Vulgaris
Keywords: azelaic acid; Clindamycin; Benzoyl peroxide; Acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; azelaic acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): A total of 110 subjects will receive clindamycin + BPO once daily in the evening for 12 weeks as per the randomization schedule.
  Interventions: Drug: Clindamycin + BPO
- Arm 2 (Experimental): A total of 110 subjects will receive azelaic acid twice daily (1 in the morning and 1 in the evening) for 12 weeks as per the randomization schedule.
  Interventions: Drug: Azelaic acid

INTERVENTIONS:
Drug: Clindamycin + BPO — Gel containing 1.2% clindamycin and 3% BPO for once daily application
  Arms: Arm 1
Drug: Azelaic acid — Cream containing 20% azelaic acid for twice daily application
  Arms: Arm 2

SUMMARY:
This is a randomized, comparator-controlled, single-blind, parallel-group study. The current study proposes to compare a fixed-dose combination product containing 3% benzoyl peroxide (BPO) and 1% clindamycin against a cream containing 20% azelaic acid for the treatment of facial acne vulgaris. The results of the study will enable a better assessment of the safety and efficacy of the new dose regime (BPO 3% + clindamycin 1%) in comparison to a well established treatment. Based on the data more evidence based recommendations will be possible to improve the treatment of subjects with acne vulgaris. A total of 220 subjects will be enrolled and will have 5 study visits (Day 1, Weeks 2, 4, 8 and 12). The duration of the study will be over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are males or females 12 to 45 years of age, inclusive.
* Subjects with acne vulgaris who have: a minimum of 17 to a maximum of 60 inflammatory facial lesions (papules and pustules), including the nose, and no more than 1 facial nodular cystic lesions and a minimum of 20 to a maximum of 125 non-inflammatory facial lesions (open and closed comedones) and an ISGA score of 2 or 3.
* Subjects agreeing not to use sun-beds or undergo any ultraviolet (UV) light treatment for 4 weeks prior to entering the study and to minimize the amount of exposure to direct sunlight for the duration of the study.
* Subjects who are capable of understanding and willing to provide signed and dated written voluntary informed consent before any protocol-specific procedures are performed. Subjects under the legal age of consent must provide assent and have the written, informed consent of both parents or legal guardians.

Exclusion Criteria:

* Unable to comply with the requirement of the study.
* Female subjects who are pregnant, breast-feeding, or sexually active and not using reliable contraception and/or not prepared to do so for the duration of the trial (a negative pregnancy test must be confirmed at Visit 1, 3, 4 and 5, for all females if menarche has occurred).
* Subjects who have any clinically relevant finding at their baseline physical examination or medical history such as severe systemic diseases or diseases of the facial skin other than acne vulgaris.
* Subjects who have facial hair that may obscure the accurate assessment of acne grade.
* Subjects who have a history or presence of regional enteritis or inflammatory bowel disease (eg, ulcerative colitis, pseudomembranous colitis, chronic diarrhea, or a history of antibiotic-associated colitis) or similar symptoms.
* Prior Therapy: Have received treatment with the following therapies at the times specified prior to Baseline: systemic retinoids [6 months]; systemic antibiotics, investigational therapy, facial procedure (chemical or laser peel, microdermabrasion, artificial UV therapy), topical corticosteroids on the face or systemic corticosteroids [4 weeks]; topical antibiotics on the face, topical anti-acne medications (eg, BPO, retinoids, azelaic acid, resorcinol, salicylates, sulfacetamide sodium and derivatives, glycolic acid) [2 weeks]; medications that are reported to exacerbate acne (eg, mega-doses of certain vitamins such as vitamin D, vitamin A, and vitamins B2, B6, and B12; haloperidol; halogens such as iodide and bromide; lithium; hydantoin; and phenobarbital) as these may impact efficacy assessments, neuromuscular blocking agents (Clindamycin has neuromuscular blocking activities, which may enhance the action of other neuromuscular blocking agents), drugs known to be photosensitizers (eg, thiazides, tetracyclines, fluoroquinolones, phenothiazines, sulfonamides) because of the possibility of increased phototoxicity [1 day].
* Subjects who are unwilling to stop using the following types of facial products during the study: astringents, toners, abradants, facials, peels containing glycolic or other acids, masks, washes or soaps containing BPO, sulfacetamide sodium or salicylic acid, non-mild facial cleansers, or moisturizers that contain retinol, salicylic acid, or alpha- or beta-hydroxy acids.
* Subjects who have a known hypersensitivity or previous allergic reaction to any of the active components (azaleic acid, lincomycin, clindamycin, BPO), or excipients of the study medication.
* Use of estrogens, including oral, implanted, and topical contraceptives, androgens, or anti-androgenic agents of less than 12 consecutive weeks prior to start of study dosing (change of the dose or drug is not permitted between 12 weeks prior study dosing until end of the study).

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 222 (Actual)
Dates: Start 2014-02-21 (Actual); Primary Completion 2014-09-08 (Actual); Study Completion 2014-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- Germany (11):
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Gilching, Bavaria
  - GSK Investigational Site, Mahlow, Brandenburg
  - GSK Investigational Site, Duelmen, Lower Saxony
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Dessau, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 200398 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200398 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200398 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200398 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200398 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200398 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200398 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 21 February 2014 to 08 September 2014 across 11 centers in Germany. A total of 222 participants were enrolled.
Pre-assignment Details: Out of 222 enrolled participants, one was assessed as screening failure and thus, 221 participants were randomized with 111 allocated to Duac and 110 to Skinoren. Four randomized participants were not treated with any study drug and therefore the intent-to-treat population consisted of 217 participants.
Groups:
- DUAC®: Participants received DUAC® (1.2 percent clindamycin + 3 percent of benzoyl peroxide [BPO]) once daily in the evening for 12 weeks as per the randomization schedule.
- SKINOREN®: Participants received SKINOREN® (20 percent azelaic acid) twice daily (1 in the morning and 1 in the evening) for 12 weeks as per the randomization schedule.
Period: Overall Study
Arm/Group | DUAC® | SKINOREN®
Started | 111 | 110
Completed | 104 | 102
Not Completed | 7 | 8
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 2 | 4
Not completed — Not in time schedule | 0 | 1
Not completed — The visit date was not in timeline | 0 | 1
Not completed — A lot of time for study for participant | 1 | 0
Not completed — Non compliance | 1 | 0

BASELINE CHARACTERISTICS:
Population: Out of 221 randomized participants, 4 participants did not receive study medication. Hence, the Intent-to-treat (ITT) population consisted of 217 participants
Groups:
- DUAC®: Participants received DUAC® (1.2 percent clindamycin and 3 percent of BPO) once daily in the evening for 12 weeks as per the randomization schedule.
- SKINOREN®: Participants received SKINOREN® (20 percent azelaic acid) twice daily (1 in the morning and 1 in the evening) for 12 weeks as per the randomization
- Total: Total of all reporting groups
Arm/Group | DUAC® | SKINOREN® | Total
Number analyzed (Participants) | 108 | 109 | 217
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.1 (7.1) | 20.0 (6.9) | 20.1 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 58 | 119
  Male | 47 | 51 | 98
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 5 | 0 | 5
  Caucasian | 94 | 102 | 196
  African | 1 | 1 | 2
  Other | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline (Day 1) of Inflammatory Lesion (IL) Count at Week 4 - Superiority Analysis
Description: A count of IL (papules and pustules, including nasal lesions) was performed at baseline and up to Week 12. Lesion counts were confined to the face. Baseline was defined at Visit 1 (Day 1). Change from Baseline in the number of IL was defined as Week 4 values minus the Baseline values. Raw data has been presented for outcome measure results; however, p value is derived from the Wilcoxon test mean scores.
Time Frame: Baseline (Day 1) and Week 4
Population: Modified intent-to-treat (MITT) population consisted of all participants in the ITT analysis set who had a baseline measurement of the number of IL and who had at least one post-baseline measurement of the number of IL.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | DUAC® | SKINOREN®
Number analyzed (Participants) | 107 | 108
Percent change | -51.9 (27.6) | -38.1 (30.9)
Statistical Analysis 1: Comparison: DUAC® vs SKINOREN®; Test type: Superiority or Other; p = 0.0004, Wilcoxon (Mann-Whitney) — Data is represented as per CTR; DUAC versus SKINOREN with a nominal alpha level of 5%, without adjustment for multiple comparisons

2. Secondary Outcome: Absolute Change From Baseline in IL, Non-inflammatory Lesions (NIL) and Calculated Total Lesions to Weeks 2, 4, 8 and 12
Description: A count of IL (papules and pustules, including nasal lesions), NIL (open and closed comedones) and total lesions was performed at baseline and up to Week 12. Lesion counts were confined to the face. Baseline was defined at Visit 1 (Day 1). Change from Baseline in the number of IL was defined as week 12 values minus the Baseline values.
Time Frame: Baseline (Day 1) up to Week 2, 4, 8, 12
Population: MITT population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | DUAC® | SKINOREN®
Number analyzed (Participants) | 107 | 108
Lesions
  IL, WEEK 2: number analyzed (Participants) | 105 | 108
  IL, WEEK 2 | -10.3 (8.3) | -6.3 (7.8)
  IL, WEEK 4: number analyzed (Participants) | 105 | 107
  IL, WEEK 4 | -14.2 (9.1) | -9.7 (8.6)
  IL, WEEK 8: number analyzed (Participants) | 104 | 102
  IL, WEEK 8 | -17.7 (9.7) | -12.7 (8.6)
  IL, WEEK 12: number analyzed (Participants) | 107 | 104
  IL, WEEK 12 | -19.6 (10.1) | -14.2 (8.9)
  NIL, WEEK 2: number analyzed (Participants) | 105 | 108
  NIL, WEEK 2 | -13.7 (19.0) | -8.5 (13.3)
  NIL, WEEK 4: number analyzed (Participants) | 105 | 107
  NIL, WEEK 4 | -21.2 (21.5) | -16.0 (19.1)
  NIL, WEEK 8: number analyzed (Participants) | 104 | 102
  NIL, WEEK 8 | -26.8 (27.1) | -20.9 (23.6)
  NIL, WEEK 12: number analyzed (Participants) | 107 | 104
  NIL, WEEK 12 | -32.0 (27.2) | -23.3 (24.9)
  Total lesion, Week 2: number analyzed (Participants) | 105 | 108
  Total lesion, Week 2 | -23.9 (22.3) | -14.8 (16.7)
  Total lesion, Week 4: number analyzed (Participants) | 105 | 107
  Total lesion, Week 4 | -35.4 (25.0) | -25.7 (22.3)
  Total lesion, Week 8: number analyzed (Participants) | 104 | 102
  Total lesion, Week 8 | -44.4 (31.3) | -33.6 (27.5)
  Total lesion, Week 12: number analyzed (Participants) | 107 | 104
  Total lesion, Week 12 | -51.6 (30.9) | -37.5 (29.0)

3. Secondary Outcome: Percentage Change From Baseline in IL, NIL and Calculated Total Lesions at Weeks 2, 4, 8 and 12
Description: A count of IL (papules and pustules, including nasal lesions),NIL (open and closed comedones) and total lesions was performed at baseline and up to Week 12. Lesion counts were confined to the face. Baseline was defined at Visit 1 (Day 1). Change from Baseline in the number of IL was defined as week 12 values minus the Baseline values.
Time Frame: Baseline (Day 1) up to Week 2, 4, 8, 12
Population: MITT population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- DUAC®: Participants received DUAC® (1.2 percent clindamycin and 3 percent of benzoyl peroxide (BPO)) once daily in the evening for 12 weeks as per the randomization schedule
Arm/Group | DUAC® | SKINOREN®
Number analyzed (Participants) | 107 | 108
Percent change
  IL, Week 2: number analyzed (Participants) | 105 | 108
  IL, Week 2 | -37.3 (27.7) | -24.2 (30.3)
  IL, Week 4: number analyzed (Participants) | 105 | 107
  IL, Week 4 | -52.2 (27.7) | -38.1 (31.1)
  IL, Week 8: number analyzed (Participants) | 104 | 102
  IL, Week 8 | -65.0 (26.3) | -49.1 (30.9)
  IL, Week 12: number analyzed (Participants) | 107 | 104
  IL, Week 12 | -72.3 (25.0) | -55.0 (29.8)
  NIL, Week 2: number analyzed (Participants) | 105 | 108
  NIL, Week 2 | -23.5 (25.3) | -14.9 (23.4)
  NIL, Week 4: number analyzed (Participants) | 105 | 107
  NIL, Week 4 | -38.1 (27.8) | -27.0 (28.2)
  NIL, Week 8: number analyzed (Participants) | 104 | 102
  NIL, Week 8 | -48.5 (39.8) | -35.5 (31.2)
  NIL, Week 12: number analyzed (Participants) | 107 | 104
  NIL, Week 12 | -60.6 (35.3) | -42.1 (37.5)
  Total lesions, Week 2: number analyzed (Participants) | 105 | 108
  Total lesions, Week 2 | -28.7 (22.3) | -18.4 (20.3)
  Total lesions, Week 4: number analyzed (Participants) | 105 | 107
  Total lesions, Week 4 | -43.8 (23.3) | -30.8 (23.0)
  Total lesions, Week 8: number analyzed (Participants) | 104 | 102
  Total lesions, Week 8 | -55.2 (30.5) | -40.1 (27.4)
  Total lesions, Week 12: number analyzed (Participants) | 107 | 104
  Total lesions, Week 12 | -64.6 (26.9) | -46.1 (31.8)

4. Secondary Outcome: Speed of Onset : Time to 50 Percent Reduction in Total Lesion Count
Description: The average time to 50 percent reduction of the calculated total lesion count was analyzed by determination of the number of days between Baseline and the first visit with a 50 percent reduction of the count.
Time Frame: Week 12
Population: MITT population. Only those participants available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | DUAC® | SKINOREN®
Number analyzed (Participants) | 91 | 60
Days | 52.0 [11.0 to 104.0] | 55.0 [12.0 to 97.0]

5. Secondary Outcome: Number of Participants With Change From Baseline in Investigator's Static Global Assessment (ISGA) to Weeks 2,4,8 and 12
Description: ISGA was conducted at all study visits. The area considered for the ISGA was confined to the face. A 0-5 point rating scale was used: 0 means Clear- Clear skin with no IL or NIL, 1 means Almost Clear- Rare NIL with no more than one small IL, 2 means Mild- Some NIL with no more than a few IL (papules/pustules only, no nodular lesions), 3 means Moderate- Up to many NIL and may have some IL, but no more than one small nodular lesion, 4 means Severe- Up to many NIL and IL, but no more than a few nodular lesions and 5 means Very Severe- Many NIL and IL and more than a few nodular lesions, may have cystic lesions.
Time Frame: Baseline (Day 1) up to Weeks 2, 4, 8, 12
Population: MITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | DUAC® | SKINOREN®
Number analyzed (Participants) | 107 | 108
Participants
  Mild (Baseline) to Almost Clear (Week 2) | 4 | 1
  Mild (Baseline) to Moderate (Week 2) | 3 | 8
  Moderate (Baseline) to Almost Clear (Week 2) | 1 | 1
  Moderate (Baseline) to Mild (Week 2) | 26 | 14
  Moderate (Baseline) to Missing (Week 2) | 2 | 0
  Mild (Baseline) to Almost Clear (Week 4) | 8 | 8
  Mild (Baseline) to Moderate (Week 4) | 1 | 4
  Mild (Baseline) to Missing (Week 4) | 0 | 1
  Moderate (Baseline) to Almost Clear (Week 4) | 11 | 3
  Moderate (Baseline) to Mild (Week 4) | 29 | 24
  Moderate (Baseline) to Severe (Week 4) | 0 | 1
  Moderate (Baseline) to Missing (Week 4) | 2 | 0
  Mild (Baseline) to Clear (Week 8) | 2 | 0
  Mild (Baseline) to Almost Clear (Week 8) | 10 | 10
  Mild (Baseline) to Moderate (Week 8) | 3 | 8
  Mild (Baseline) to Missing (Week 8) | 0 | 4
  Moderate (Baseline) to Clear (Week 8) | 1 | 0
  Moderate (Baseline) to Almost Clear (Week 8) | 15 | 5
  Moderate (Baseline) To Mild (Week 8) | 32 | 27
  Moderate (Baseline) to Missing (Week 8) | 3 | 2
  Mild (Baseline) to Clear (Week 12) | 3 | 1
  Mild (Baseline) to Almost Clear (Week 12) | 12 | 9
  Mild (Baseline) to Moderate (Week 12) | 2 | 8
  Mild (Baseline) to Missing (Week 12) | 0 | 2
  Moderate (Baseline) to Clear (Week 12) | 2 | 0
  Moderate (Baseline) to Almost Clear (Week 12) | 19 | 9
  Moderate (Baseline) to Mild (Week 12) | 33 | 26
  Moderate (Baseline) to Severe (Week 12) | 0 | 2
  Moderate (Baseline) to Missing (Week 12) | 0 | 2

6. Secondary Outcome: Number of Participants With Change From Baseline in Local Tolerability as Per Investigator's Assessment at Weeks 2,4,8,12
Description: Tolerability was assessed by investigator on a 0-3 point rating scale for erythema (0- None, 1- Slight, 2- Some and 3- Very red), dryness (0- None, 1- Slight, 2- Some and 3- Very dry) and peeling (0- None, 1- Slight, 2- Moderate and 3- Strong). A shift table was provided to deduce how the results are varying from the baseline visit to post-baseline visits. Change from Baseline is the value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1) and Weeks 2, 4, 8, 12
Population: MITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | DUAC® | SKINOREN®
Number analyzed (Participants) | 107 | 108
Participants
  Erythema None (Baseline) To Slight (Week 2) | 11 | 18
  Erythema None (Baseline) To Some (Week 2) | 0 | 1
  Erythema None (Baseline) To Missing (Week 2) | 1 | 0
  Erythema Slight (Basline) To None (Week 2) | 12 | 12
  Erythema Slight (Baseline) To Some (Week 2) | 1 | 8
  Erythema Slight (Baseline) To Missing (Week 2) | 1 | 0
  Erythema Some (Baseline) To None (Week 2) | 3 | 1
  Erythema Some (Baseline) To Slight (Week 2) | 10 | 11
  Erythema Very Red (Baseline) To Slight (Week 2) | 1 | 1
  Erythema Very Red (Baseline) To Some (Week 2) | 2 | 2
  Erythema Missing (Baseline) To None (Week 2) | 1 | 0
  Erythema None (Baseline) To Slight (Week 4) | 9 | 13
  Erythema None (Baseline) To Some (Week 4) | 1 | 3
  Erythema None (Baseline) To Missing (Week 4) | 1 | 0
  Erythema Slight (Baseline) To None (Week 4) | 18 | 19
  Erythema Slight (Baseline) To Some (Week 4) | 3 | 1
  Erythema Slight (Baseline) To Missing (Week 4) | 1 | 1
  Erythema Some (Baseline) To None (Week 4) | 5 | 3
  Erythema Some (Baseline) To Slight (Week 4) | 11 | 9
  Erythema Some (Baseline) To Missing (Week 4) | 0 | 1
  Erythema Very Red (Baseline) To Slight (Week 4) | 2 | 2
  Erythema Very Red (Baseline) To Some (Week 4) | 1 | 1
  Erythema Missing (Baseline) To None (Week 4) | 1 | 0
  Erythema None (Baseline) To Slight (Week 8) | 10 | 19
  Erythema None (Baseline) To Some (Week 8) | 0 | 2
  Erythema None (Baseline) To Missing (Week 8) | 1 | 2
  Erythema Slight (Baseline) To None (Week 8) | 15 | 17
  Erythema Slight (Baseline) To Some (Week 8) | 5 | 1
  Erythema Slight (Baseline) To Missing (Week 8) | 2 | 3
  Erythema Some (Baseline) To None (Week 8) | 8 | 1
  Erythema Some (Baseline) To Slight (Week 8) | 9 | 12
  Erythema Some (Baseline) To Very Red (Week 8) | 1 | 0
  Erythema Some (Baseline) To Missing (Week 8) | 0 | 1
  Erythema Very Red (Baseline) To None (Week 8) | 2 | 0
  Erythema Very Red (Baseline) To Slight (Week 8) | 1 | 3
  Erythema Missing (Baseline) To Slight (Week 8) | 1 | 0
  Erythema None (Baseline) To Slight (Week 12) | 6 | 18
  Erythema None (Baseline) To Missing (Week 12) | 0 | 2
  Erythema Slight (Baseline) To None (Week 12) | 21 | 22
  Erythema Slight (Baseline) To Some (Week 12) | 0 | 2
  Erythema Slight (Baseline) To Very Red (Week 8) | 1 | 0
  Erythema Slight (Baseline) To Missing (Week 12) | 0 | 1
  Erythema Some (Baseline) To None (Week 12) | 9 | 4
  Erythema Some (Baseline) To Slight (Week 12) | 8 | 9
  Erythema Some (Baseline) To Missing (Week 12) | 0 | 1
  Erythema Very Red (Baseline) To None (Week 12) | 0 | 2
  Erythema Very Red (Baseline) To Slight (Week 12) | 1 | 1
  Erythema Missing (Baseline) To Slight (Week 12) | 1 | 0
  Peeling None (Baseline) To Slight (Week 2) | 13 | 11
  Peeling None (Baseline) To Moderate (Week 2) | 1 | 0
  Peeling None (Baseline) To Missing (Week 2) | 2 | 0
  Peeling Slight (Baseline) To None (Week 2) | 8 | 8
  Peeling Slight (Baseline) To Moderate (Week 2) | 3 | 2
  Peeling Moderate (Baseline) To None (Week 2) | 2 | 0
  Peeling Moderate (Baseline) To Slight (Week 2) | 2 | 1
  Peeling Missing (Baseline) To None (Week 2) | 1 | 0
  Peeling None (Baseline) To Slight (Week 4) | 9 | 11
  Peeling None (Baseline) To Missing (Week 4) | 2 | 1
  Peeling Slight (Baseline) To None (Week 4) | 15 | 13
  Peeling Slight (Baseline) To Moderate (Week 4) | 1 | 1
  Peeling Moderate (Baseline) To None (Week 4) | 2 | 1
  Peeling Moderate (Baseline) To Slight (Week 4) | 1 | 0
  Peeling Missing (Baseline) To None (Week 4) | 1 | 0
  Peeling None (Baseline) To Slight (Week 8) | 9 | 10
  Peeling None (Baseline) To Missing (Week 8) | 3 | 5
  Peeling Slight (Baseline) To None (Week 8) | 18 | 12
  Peeling Slight (Baseline) To Missing (Week 8) | 0 | 1
  Peeling Moderate (Baseline) To None (Week 8) | 3 | 1
  Peeling Moderate (Baseline) To Slight (Week 8) | 1 | 0
  Peeling Missing (Baseline) To None (Week 8) | 1 | 0
  Peeling None (Baseline) To Slight (Week 12) | 7 | 11
  Peeling None (Baseline) To Missing (Week 12) | 0 | 3
  Peeling Slight (Baseline) To None (Week 12) | 14 | 15
  Peeling Slight (Baseline) To Missing (Week 12) | 0 | 1
  Peeling Moderate (Baseline) To None (Week 12) | 2 | 0
  Peeling Moderate (Baseline) To Slight (Week 12) | 2 | 1
  Peeling Missing (Baseline) To None (Week 12) | 1 | 0
  Dryness None (Baseline) To Slight (Week 2) | 14 | 9
  Dryness None (Baseline) To Some (Week 2) | 1 | 3
  Dryness None (Baseline) To Missing (Week 2) | 2 | 0
  Dryness Slight (Baseline) To None (Week 2) | 11 | 7
  Dryness Slight (Baseline) To Some (Week 2) | 3 | 6
  Dryness Some (Baseline) To None (Week 2) | 4 | 2
  Dryness Some (Baseline) To Slight (Week 2) | 1 | 2
  Dryness Missing (Baseline) To None (Week 2) | 1 | 0
  Dryness None (Baseline) To Slight (Week 4) | 9 | 12
  Dryness None (Baseline) To Missing (Week 4) | 2 | 1
  Dryness Slight (Baseline) To None (Week 4) | 14 | 10
  Dryness Slight (Baseline) To Some (Week 4) | 2 | 3
  Dryness Some (Baseline) To None (Week 4) | 4 | 1
  Dryness Some (Baseline) To Slight (Week 4) | 3 | 5
  Dryness Missing (Baseline) To None (Week 4) | 1 | 0
  Dryness None (Baseline) To Slight (Week 8) | 8 | 11
  Dryness None (Baseline) To Missing (Week 8) | 3 | 5
  Dryness Slight (Baseline) To None (Week 8) | 19 | 12
  Dryness Slight (Baseline) To Some (Week 8) | 0 | 1
  Dryness Slight (Baseline) To Missing (Week 8) | 0 | 1
  Dryness Some (Baseline) To None (Week 8) | 5 | 1
  Dryness Some (Baseline) To Slight (Week 8) | 4 | 5
  Dryness Missing (Baseline) To None (Week 8) | 1 | 0
  Dryness None (Baseline) To Some (Week 12) | 1 | 0
  Dryness None (Baseline) To Slight (Week 12) | 2 | 8
  Dryness None (Baseline) To Missing (Week 12) | 0 | 3
  Dryness Slight (Baseline) To None (Week 12) | 14 | 15
  Dryness Slight (Baseline) To Some (Week 12) | 0 | 1
  Dryness Slight (Baseline) To Missing (Week 12) | 0 | 1
  Dryness Some (Baseline) To None (Week 12) | 6 | 3
  Dryness Some (Baseline) To Slight (Week 12) | 3 | 3
  Dryness Missing (Baseline) To None (Week 12) | 1 | 0

7. Secondary Outcome: Number of Participants With Participant Global Change Assessment Score 12 Weeks
Description: An SGCA was conducted by the participant to assess the efficacy of treatment on Week 2, 4, 8 and 12 as Very Much Improved, Much Improved, Minimally Improved, No Change, Minimally Worse, Much Worse, Very Much Worse and missing.
Time Frame: Weeks 2, 4, 8 and 12
Population: MITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | DUAC® | SKINOREN®
Number analyzed (Participants) | 107 | 108
Participants
  Very much improved (Week 2) | 4 | 2
  Much improved (Week 2) | 51 | 30
  Minimally improved (Week 2) | 44 | 56
  No change (Week 2) | 6 | 14
  Minimally worse (Week 2) | 0 | 6
  Missing (Week 2) | 2 | 0
  Very much improved (Week 4) | 5 | 0
  Much improved (Week 4) | 48 | 39
  Minimally improved (Week 4) | 44 | 49
  No change (Week 4) | 2 | 12
  Minimally worse (Week 4) | 6 | 7
  Missing (Week 4) | 2 | 1
  Very much improved (Week 8) | 9 | 1
  Much improved (Week 8) | 54 | 44
  Minimally improved (Week 8) | 30 | 32
  No change (Week 8) | 7 | 15
  Minimally worse (Week 8) | 3 | 8
  Much worse (Week 8) | 1 | 1
  Very much worse (Week 8) | 0 | 1
  Missing (Week 8) | 3 | 6
  Very much improved (Week 12) | 14 | 8
  Much improved (Week 12) | 48 | 38
  Minimally improved (Week 12) | 29 | 33
  No change (Week 12) | 10 | 17
  Minimally worse (Week 12) | 4 | 5
  Much worse (Week 12) | 0 | 2
  Very much worse (Week 12) | 2 | 1
  Missing (Week 12) | 0 | 4

8. Secondary Outcome: Number of Participants With Change From Baseline in Local Tolerability as Per Participant's Assessment at Weeks 2, 4, 8 and 12
Description: Tolerability was assessed by the participants based on a 0-3 point rating scale for stinging/burning (S/B) and pruritus of the face (0- None, 1- Slight, 2- Moderate and 3- Strong). A shift table was provided to deduce how the results are varying from the Baseline visit to post-baseline visits.
Time Frame: Baseline (Day 1), Weeks 2, 4, 8 and 12
Population: MITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | DUAC® | SKINOREN®
Number analyzed (Participants) | 107 | 108
Participants
  S/B None (Baseline) To Slight (Week 2) | 14 | 23
  S/B None (Baseline) To Moderate (Week 2) | 4 | 8
  S/B None (Baseline) To Strong (Week 2) | 1 | 4
  S/B None (Baseline) To Missing (Week 2) | 2 | 0
  S/B Slight (Baseline) To None (Week 2) | 14 | 10
  S/B Slight (Baseline) To Moderate (Week 2) | 3 | 2
  S/B Slight (Baseline) To Strong (Week 2) | 0 | 2
  S/B Moderate (Baseline) To None (Week 2) | 0 | 1
  S/B Moderate (Baseline) To Slight (Week 2) | 1 | 3
  S/B Strong (Baseline) To None (Week 2) | 0 | 1
  S/B Missing (Baseline) To None (Week 2) | 1 | 0
  S/B None (Baseline) To Slight (Week 4) | 11 | 29
  S/B None (Baseline) To Moderate (Week 4) | 1 | 6
  S/B None (Baseline) To Missing (Week 4) | 2 | 1
  S/B Slight (Baseline) To None (Week 4) | 12 | 9
  S/B Slight (Baseline) To Moderate (Week 4) | 1 | 1
  S/B Slight (Baseline) To Strong (Week 4) | 0 | 1
  S/B Moderate (Baseline) To None (Week 4) | 0 | 2
  S/B Moderate (Baseline) To Slight (Week 4) | 1 | 3
  S/B Moderate (Baseline) To Strong (Week 4) | 0 | 1
  S/B Strong (Baseline) To None (Week 4) | 0 | 1
  S/B Missing (Baseline) To Slight (Week 4) | 1 | 0
  S/B None (Baseline) To Slight (Week 8) | 5 | 21
  S/B None (Baseline) To Moderate (Week 8) | 1 | 4
  S/B None (Baseline) To Missing (Week 8) | 3 | 5
  S/B None (Baseline) To Strong (Week 8) | 0 | 1
  S/B Slight (Baseline) To None (Week 8) | 18 | 10
  S/B Slight (Baseline) To Moderate (Week 8) | 1 | 1
  S/B Slight (Baseline) To Strong (Week 8) | 0 | 1
  S/B Moderate (Baseline) To None (Week 8) | 0 | 1
  S/B Moderate (Baseline) To Slight (Week 8) | 1 | 2
  S/B Moderate (Baseline) To Missing (Week 8) | 0 | 1
  S/B Strong (Baseline) To None (Week 8) | 0 | 1
  S/B Missing (Baseline) To None (Week 8) | 1 | 0
  S/B None (Baseline) To Slight (Week 12) | 6 | 19
  S/B None (Baseline) To Moderate (Week 12) | 1 | 5
  S/B None (Baseline) To Strong (Week 12) | 1 | 2
  S/B None (Baseline) To Missing (Week 12) | 1 | 4
  S/B Slight (Baseline) To None (Week 12) | 18 | 9
  S/B Slight (Baseline) To Moderate (Week 12) | 0 | 3
  S/B Slight (Baseline) To Strong (Week 12) | 0 | 1
  S/B Moderate (Baseline) To None (Week 12) | 1 | 2
  S/B Moderate (Baseline) To Slight (Week 12) | 0 | 3
  S/B Strong (Baseline) To Slight (Week 12) | 0 | 1
  S/B Missing (Baseline) To None (Week 12) | 1 | 0
  Pruritus None (Baseline) To Slight (Week 2) | 14 | 27
  Pruritus None (Baseline) To Moderate (Week 2) | 4 | 7
  Pruritus None (Baseline) To Strong (Week 2) | 0 | 1
  Pruritus None (Baseline) To Missing (Week 2) | 2 | 0
  Pruritus Slight (Baseline) To None (Week 2) | 13 | 10
  Pruritus Slight (Baseline) To Moderate (Week 2) | 5 | 9
  Pruritus Slight (Baseline) To Strong (Week 2) | 1 | 4
  Pruritus Moderate (Baseline) To None (Week 2) | 2 | 4
  Pruritus Moderate (Baseline) To Slight (Week 2) | 1 | 1
  Pruritus Missing (Baseline) To None (Week 2) | 1 | 0
  Pruritus None (Baseline) To Slight (Week 4) | 14 | 30
  Pruritus None (Baseline) To Moderate (Week 4) | 2 | 5
  Pruritus None (Baseline) To Missing (Week 4) | 2 | 1
  Pruritus Slight (Baseline) To None (Week 4) | 17 | 12
  Pruritus Slight (Baseline) To Moderate (Week 4) | 2 | 6
  Pruritus Slight (Baseline) To Strong (Week 4) | 0 | 1
  Pruritus Moderate (Baseline) To None (Week 4) | 2 | 2
  Pruritus Moderate (Baseline) To Slight (Week 4) | 2 | 2
  Pruritus Missing (Baseline) To None (Week 4) | 1 | 0
  Pruritus None (Baseline) To Slight (Week 8) | 13 | 26
  Pruritus None (Baseline) To Missing (Week 8) | 3 | 3
  Pruritus None (Baseline) To Strong (Week 8) | 0 | 1
  Pruritus Slight (Baseline) To None (Week 8) | 21 | 11
  Pruritus Slight (Baseline) To Moderate (Week 8) | 4 | 4
  Pruritus Slight (Baseline) To Strong (Week 8) | 0 | 2
  Pruritus Slight (Baseline) To Missing (Week 8) | 0 | 3
  Pruritus Moderate (Baseline) To None (Week 8) | 3 | 2
  Pruritus Moderate (Baseline) To Slight (Week 8) | 1 | 3
  Pruritus Strong (Baseline) To Moderate (Week 8) | 0 | 1
  Pruritus Missing (Baseline) To None (Week 8) | 1 | 0
  Pruritus None (Baseline) To Slight (Week 12) | 11 | 22
  Pruritus None (Baseline) To Moderate (Week 12) | 1 | 3
  Pruritus None (Baseline) To Strong (Week 12) | 0 | 1
  Pruritus None (Baseline) To Missing (Week 12) | 0 | 4
  Pruritus Slight (Baseline) To None (Week 12) | 22 | 11
  Pruritus Slight (Baseline) To Moderate (Week 12) | 2 | 6
  Pruritus Slight (Baseline) To Strong (Week 12) | 0 | 2
  Pruritus Moderate (Baseline) To None (Week 12) | 3 | 1
  Pruritus Moderate (Baseline) To Slight (Week 12) | 1 | 4
  Pruritus Strong (Baseline) To Slight (Week 12) | 0 | 1
  Pruritus Missing (Baseline) To None (Week 12) | 1 | 0

9. Secondary Outcome: Number of Participants With Participant Satisfaction Score at Week 12 (Simple Grading)
Description: The product acceptability and preference questionnaire (PAP-Q ) served as a patient satisfaction score and was performed only once at the final study visit (ie, after 12 weeks (V5) or earlier in case of premature termination). Severity of each facial acne sign and symptom (scaling, redness, dryness, burning, itching) was based on a 0-5 point rating scale (0- None, 1- Very minimal, 2- Mild, 3- Moderate, 4- Severe, 5- Very severe).
Time Frame: Week 12
Population: MITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | DUAC® | SKINOREN®
Number analyzed (Participants) | 107 | 108
Participants
  Redness, None | 55 | 47
  Redness, Very minimal | 32 | 20
  Redness, Mild | 8 | 17
  Redness, Moderate | 9 | 13
  Redness, Severe | 2 | 5
  Redness, Very severe | 1 | 2
  Redness, Not applicable | 0 | 1
  Dryness, None | 43 | 41
  Dryness, Very minimal | 32 | 28
  Dryness, Mild | 20 | 24
  Dryness, Moderate | 9 | 7
  Dryness, Severe | 2 | 2
  Dryness, Very severe | 1 | 2
  Dryness, Not applicable | 0 | 1
  Burning, None | 90 | 50
  Burning, Very minimal | 8 | 28
  Burning, Mild | 5 | 12
  Burning, Moderate | 3 | 9
  Burning, Severe | 1 | 5
  Burning, Very severe | 0 | 0
  Burning, Not applicable | 0 | 1
  Itching, None | 73 | 38
  Itching, Very minimal | 17 | 30
  Itching, Mild | 10 | 20
  Itching, Moderate | 6 | 11
  Itching, Severe | 1 | 3
  Itching, Very severe | 0 | 2
  Itching, Not applicable | 0 | 1
  Scaling, None | 69 | 77
  Scaling, Very minimal | 24 | 9
  Scaling, Mild | 7 | 7
  Scaling, Moderate | 2 | 7
  Scaling, Severe | 4 | 4
  Scaling, Very severe | 1 | 0
  Scaling, Not applicable | 0 | 1

10. Secondary Outcome: Number of Treatment Adherent Participants at Week 12
Description: The general assessment of 'overall satisfaction' with study therapy was assessed at week 12 on a 0-4 point rating scale (0-Very satisfied, 1- Satisfied, 2- Neutral, 3- Unsatisfied and 4- Very unsatisfied).
Time Frame: Week 12
Population: MITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | DUAC® | SKINOREN®
Number analyzed (Participants) | 107 | 108
Participants
  Very satisfied | 41 | 26
  Satisfied | 61 | 43
  Neutral | 4 | 21
  Unsatisfied | 1 | 11
  Very unsatisfied | 0 | 3

11. Secondary Outcome: Absolute Change From Baseline in Total Score as Per Dermatology Life Quality Index (DLQI) at Week 2,4,8 and 12
Description: This outcome measure was a measure of quality of life (QOL). The DLQI was used to assess the quality of life at each visit. Participants completed the questionnaire to evaluate how their acne has affected their life. The DLQI is a 10 item questionnaire, which addresses feelings, daily activities, leisure, work, school, personal relationships, and treatment. Each question was scored out of 0-3, as follows: 0- Not at all, 1- A little, 2- A lot, 3- very much, indicating 0 as the least and 3 as the best quality Index. The sub-scale scores of 10 questions were combined and a composite score was presented. The total score ranged from 0 to 30, 0 indicated the least and highest score indicated the best quality Index. The DLQI was for participants with 17 to 45 years of age. Baseline was defined at Visit 1 (Day 1). Change from Baseline is the value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1) up to Weeks 2, 4, 8, 12
Population: MITT population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DUAC® | SKINOREN®
Number analyzed (Participants) | 62 | 61
Scores on a scale
  Week 2: number analyzed (Participants) | 54 | 53
  Week 2 | -2.28 (2.81) | -2.17 (3.72)
  Week 4: number analyzed (Participants) | 56 | 52
  Week 4 | -3.39 (3.33) | -3.15 (3.52)
  Week 8: number analyzed (Participants) | 55 | 50
  Week 8 | -4.04 (3.70) | -3.38 (4.60)
  Week 12: number analyzed (Participants) | 57 | 51
  Week 12 | -4.46 (3.80) | -3.12 (4.94)

12. Secondary Outcome: Absolute Change From Baseline in Total Score as Per Children's Dermatology Life Quality Index (CDLQI) at Week 2,4,8 and 12
Description: This outcome measure was a measure of QOL. The CDLQI was used to assess the quality of life at each visit. Participants completed the questionnaire to evaluate how their acne has affected their life. The DLQI is a 10 item questionnaire, which addresses feelings, daily activities, leisure, work, school, personal relationships, and treatment. Each question was scored out of 0-3, as follows: 0- Not at all, 1- A little, 2- A lot, 3- very much, indicating 0 as the least and 3 as the best quality Index. The sub-scale scores of 10 questions were combined and a composite score was presented. The total score ranged from 0 to 30, 0 indicated the least and highest score indicated the best quality Index. The CDLQI was for participants with 12 to 16 years of age. Baseline was defined at Visit 1 (Day 1). Change from Baseline is the value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1) up to Weeks 2, 4, 8, 12
Population: MITT population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DUAC® | SKINOREN®
Number analyzed (Participants) | 38 | 42
Scores on a scale
  Week 2 | -2.61 (2.89) | -1.31 (2.29)
  Week 4 | -2.55 (2.41) | -1.55 (2.01)
  Week 8 | -2.68 (2.76) | -1.67 (2.34)
  Week 12 | -2.87 (2.75) | -1.55 (2.56)

13. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (TESAEs) Related to Study Medication
Description: Adverse events are defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Serious adverse events are defined as any untoward medical occurrence that results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect and medically significant. TEAEs and TESAEs were reported up to 12 weeks.
Time Frame: Up to Week 12
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | DUAC® | SKINOREN®
Number analyzed (Participants) | 108 | 109
Participants
  TEAE | 60 | 76
  TESAE | 2 | 3
  TEAEs related to the study drug | 15 | 36
  TESAEs related to the study drug | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected up to Week 12.
Description: Intent-to-treat population consisted of all participants who were randomized and who used the test medication at least once.
Arm/Group | DUAC® | SKINOREN®
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/109
Serious Adverse Events (participants affected / at risk) | 2/108 | 3/109
Other Adverse Events (participants affected / at risk) | 32/108 | 55/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DUAC® (N=108) | SKINOREN® (N=109)
Brucellosis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Stress (Psychiatric disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Vulval haematoma (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DUAC® (N=108) | SKINOREN® (N=109)
Application site pain (General disorders) | 7 | 22
Application site pruritus (General disorders) | 8 | 25
Nasopharyngitis (Infections and infestations) | 10 | 20
Headache (Nervous system disorders) | 16 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.